CLINICAL TRIAL: NCT06752161
Title: Urinary Tract Infections in Patients with Threatened Preterm Labor
Brief Title: Urinary Infection in Pregnant Women with Urinary Infection
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Gamal M.fekry, Lecturer of obstetric and gynecology, specialist of Uro gynecology, Assiut University
Other Study IDs: UTIP
Record Dates: First submitted 2024-12-20; First posted 2024-12-30 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-12

CONDITIONS: Threatened Preterm Labour
Keywords: UTI; Preterm labour
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Urinalysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pregnant women with threatened preterm labour: Patients with UTI and preterm labour
  Interventions: Other: Urine analysis

INTERVENTIONS:
Other: Urine analysis — Urine analysis and culture for Screening and diagnostic tools for UTI in pregnant women

SUMMARY:
Urine analysis and culture in patients with threatened preterm labour

DETAILED DESCRIPTION:
UTI is an infection of the kidneys, bladder, or urethra. Infectious cystitis is the most common type of UTI, which is caused by a bacterial infection of the bladder. Lifetime incidence of UTIs is 50% to 60% in adult women.UTIs are among the most common conditions encountered in primary care, hospitals, and extended care facilities . Total direct costs of UTI treatment (without cultures) have been estimated at US $25.5 billion annually.Despite an exceptionally high prevalence of bacteriuria in the population, these infections rarely cause significant renal damage.Sexual intercourse is the strongest risk factor. Any lifetime sexual activity and any sexual activity during the past year are strongly associated with recurrent UTI. Even the relatively small amounts of spermicide coating condoms increases the risk of UTI. Post-menopausal absence of oestrogen is a risk factor for UTIs. Topical oestrogen reduces UTIs in post-menopausal women; Oestrogenisation of the vaginal mucosa promotes lactobacilli colonisation, which reduces the presence of uropathogens and thus the risk of UTIs and is not recommended over the use of topical oestrogen therapy. Urinary incontinence and oestrogen supplementation have also been associated with UTI in older women, although the reasons for this are incompletely understood. positive family history of UTIs is associated with a two- to fourfold increase in risk of recurrent UTI . Bacteriuria occurs in the presence of indwelling or intermittent catheters, and asymptomatic bacteriuria does not require treatment. Gestational and pregestational diabetes are considered a more predominant risk factor in older women.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with preterm labor

Exclusion Criteria:

* renal disease Intrauterine fetal death

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with threatened preterm labor
Sampling Method: Non-Probability Sample
Enrollment: 224 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
percent of urinary tract infections in threatened preterm labor | 1 month
  Percentage of women with threatened preterm labor diagnosed with urinary tract infection

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Seif al nasr, MBBCH, Principal Investigator — Women's Health Hospital Resident
Locations (1):
- Women's Health Hospital, Asyut, Egypt